CLINICAL TRIAL: NCT07389577
Title: A Randomized, Double-masked, Multicenter, Parallel Group, Phase 3 Clinical Trial to Compare the Efficacy and Safety of JL14002 Monoclonal Antibody Injection Versus Ranibizumab Injection in Patients With Neovascular (Wet) Age-Related Macular Degeneration (wAMD)
Brief Title: A Study to Compare JL14002 to Lucentis® in Subjects With Wet Age-related Macular Degeneration (wAMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jecho Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JechoBiopharm; CTR20213179 (Other: Center For Drug Evaluation, National Medical Products Administration, China)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Phase3; wAMD; Ranibizumab; Lucentis
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JL14002 Experimental Arm(Drug: JL14002 monoclonal antibody) (Experimental): For the first 12 weeks, a fixed dosing regimen will be administered, consisting of 0.5 mg JL14002 once every 4 weeks for a total of 3 consecutive doses. From Week 12 through Week 48, treatment will transition to a pro re nata (PRN) regimen based on pre-specified retreatment criteria.
  Interventions: Drug: JL14002 monoclonal antibody(Fixed dosing regimen); Drug: JL14002 monoclonal antibody(PRN)
- Active Comparator Arm 1 (Drug: Ranibizumab→JL14002 monoclonal antibody) (Active Comparator): For the first 12 weeks, a fixed dosing regimen will be administered, consisting of 0.5 mg Ranibizumab once every 4 weeks for a total of 3 consecutive doses. From Week 12 through Week 48, treatment will transition to a pro re nata (PRN) regimen based on pre-specified retreatment criteria., subjects will receive the JL14002 treatment
  Interventions: Drug: JL14002 monoclonal antibody(Fixed dosing regimen); Drug: JL14002 monoclonal antibody(PRN)
- Active Comparator Arm 2 (Drug:Ranibizumab) (Active Comparator): For the first 12 weeks, a fixed dosing regimen will be administered, consisting of 0.5 mg Ranibizumab once every 4 weeks for a total of 3 consecutive doses. From Week 12 through Week 48, treatment will transition to a pro re nata (PRN) regimen based on pre-specified retreatment criteria.
  Interventions: Drug: Ranibizumab(Fixed dosing regimen); Drug: Ranibizumab(PRN)

INTERVENTIONS:
Drug: JL14002 monoclonal antibody(Fixed dosing regimen) — For the first 12 weeks, a fixed dosing regimen will be administered, consisting of 0.5 mg JL14002 once every 4 weeks for a total of 3 consecutive doses.
  Other Names: Intravitreal (IVT) injection
  Arms: Active Comparator Arm 1 (Drug: Ranibizumab→JL14002 monoclonal antibody); JL14002 Experimental Arm(Drug: JL14002 monoclonal antibody)
Drug: Ranibizumab(Fixed dosing regimen) — For the first 12 weeks, a fixed dosing regimen will be administered, consisting of 0.5 mg Ranibizumab once every 4 weeks for a total of 3 consecutive doses.
  Other Names: Intravitreal (IVT) injection
  Arms: Active Comparator Arm 2 (Drug:Ranibizumab)
Drug: JL14002 monoclonal antibody(PRN) — From Week 12 through Week 48, treatment will transition to a pro re nata (PRN) regimen. Patients will receive 0.5 mg of JL14002 monoclonal antibody injection as needed, based on pre-specified retreatment criteria.
  Other Names: Intravitreal (IVT) injection; pro re nata (PRN)
  Arms: Active Comparator Arm 1 (Drug: Ranibizumab→JL14002 monoclonal antibody); JL14002 Experimental Arm(Drug: JL14002 monoclonal antibody)
Drug: Ranibizumab(PRN) — From Week 12 through Week 48, treatment will transition to a pro re nata (PRN) regimen. Patients will receive 0.5 mg of Ranibizumab injection as needed, based on pre-specified retreatment criteria.
  Other Names: Intravitreal (IVT) injection; pro re nata (PRN)
  Arms: Active Comparator Arm 2 (Drug:Ranibizumab)

SUMMARY:
This is a randomised, double-masked, parallel group, multicentre study to evaluate the efficacy and safety of JL14002 compared to Lucentis® in subjects with wAMD.

DETAILED DESCRIPTION:
Subjects will be randomised in a 2:1:1 ratio into the JL14002 Experimental Arm, Active Comparator Arm 1, and Active Comparator Arm 2. During the first 12 weeks, all subjects will receive fixed dosing at intervals of every 4 weeks (0.5 mg per dose), with a total of three consecutive doses. Subjects in the JL14002 experimental arm will receive JL14002 monoclonal antibody injection, while those in active comparator arm 1 and active comparator arm 2 will receive ranibizumab injection. Starting from week 12, all subjects will transition to a pro re nata (PRN) dosing regimen. Based on the PRN criteria assessed by the investigator, subjects in the JL14002 experimental arm and active comparator arm 1 will receive JL14002 monoclonal antibody injection as needed, while subjects in active comparator arm 2 will receive ranibizumab injection as needed. All subjects will be required to return to the study site every 4 weeks for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

1.Ability to understand and voluntarily sign the informed consent form, and willingness to comply with all trial protocol-specified follow-up visits.

2.Aged 50 to 80 years (inclusive), male or female. 3.The study eye must meet all the following criteria:

1. Diagnosis of wet Age-related Macular Degeneration (wAMD) with active disease at screening, defined by the presence of ≥1 of the following macular lesions:a) Intraretinal fluid; b) Intraretinal lipid exudation or subretinal fluid; c) Subretinal fluid; d) Subretinal hemorrhage; e) Retinal pigment epithelial detachment (PED).
2. Best Corrected Visual Acuity (BCVA) score between 75 and 24 letters (inclusive) as measured by ETDRS chart at screening (Snellen equivalent: 20/32 to 20/320).

Exclusion Criteria:

1. Previous treatment with photodynamic therapy (PDT) or any combination therapy involving PDT in either eye.
2. Any intravitreal anti-VEGF therapy (e.g., bevacizumab, aflibercept, ranibizumab, conbercept) in either eye within 90 days before the first dose.
3. Previous ocular surgery in the study eye, including but not limited to: macular translocation, glaucoma filtration surgery, subfoveal laser photocoagulation, vitrectomy, transpupillary thermotherapy, or any other surgery for AMD.
4. Subretinal hemorrhage in the study eye involving the fovea, with an area ≥4 disc areas (DA) on FFA.
5. Presence of subfoveal fibrosis, scar, geographic atrophy, or dense subfoveal hard exudates in the study eye.
6. Choroidal neovascularization (CNV) in the study eye due to causes other than wAMD (e.g., ocular histoplasmosis, pathologic myopia, angioid streaks, trauma).
7. Any concurrent ocular disease (other than wAMD) or history thereof in the study eye that could confound assessment of the macula or central vision (e.g., diabetic retinopathy, retinal vein occlusion, central serous chorioretinopathy, macular hole, epiretinal membrane, vitreomacular traction).
8. Any ocular condition in the study eye that, per investigator judgment, may require treatment during the study, lead to vision loss, or preclude adequate fundus imaging/assessment (e.g., significant media opacity, pupillary miosis).
9. Intraocular or periocular surgery in the study eye within 90 days before the first dose (excluding uncomplicated eyelid surgery >28 days prior). Parafoveal laser or cataract surgery within this period is excluded.
10. History of corneal transplantation in the study eye.
11. Active intraocular, extraocular, or periocular inflammation in either eye at screening.
12. Active ocular infection in either eye at screening (e.g., conjunctivitis, keratitis, scleritis, endophthalmitis, uveitis).
13. History of idiopathic or autoimmune-associated uveitis in either eye.
14. Current vitreous hemorrhage in the study eye or history thereof within 28 days before the first dose.
15. Aphakia (excluding pseudophakia) or rupture of the posterior lens capsule in the study eye (except status post YAG laser capsulotomy).
16. Advanced glaucoma or optic neuropathy involving/threatening the central visual field in the study eye; or uncontrolled intraocular pressure (IOP ≥25 mmHg despite treatment).
17. High myopia (spherical equivalent ≤ -6 diopters) in the study eye.
18. Current or anticipated use of medications with known retinal, lens, or optic nerve toxicity (e.g., chloroquine/hydroxychloroquine, ethambutol, tamoxifen, phenothiazines).
19. History of severe allergic reaction to biologics, or known hypersensitivity to JL14002, ranibizumab, fluorescein/ICG, mydriatics, or related topical agents.
20. Active systemic infection requiring therapy.
21. Poorly controlled autoimmune disease.
22. Any condition that, per investigator judgment, poses a high risk for complications or confounds results (e.g., uncontrolled hypertension [SBP≥160 or DBP≥100 mmHg], HbA1c ≥8%).
23. Recent corticosteroid use meeting any of the following:

1) Study eye (intraocular/subconjunctival): Intermediate-/short-acting (e.g., triamcinolone) within 90 days; long-acting/sustained-release (e.g., dexamethasone implant) within 180 days.

2) Study eye (periocular): Injection within 28 days before screening; topical ocular use for ≥30 continuous days within 90 days.

3) Systemic: Within 5 days before screening or anticipated need during study (excluding topical, inhaled, intranasal, intra-articular, or short-term oral [<2 weeks] use).

24.Fellow eye BCVA <24 letters (Snellen <20/320) or presence of other potentially blinding conditions.

25.Systemic anti-VEGF therapy within 90 days before the first dose. 26.History of malignancy within 5 years (exceptions: adequately treated basal/squamous cell skin cancer, carcinoma in situ of cervix/breast).

27.Clinically significant abnormal liver or renal function:1) ALT or AST ≥2 × ULN;2) Creatinine or BUN ≥1.5 × ULN 28.Coagulopathy (PT ≥ ULN +3 sec; aPTT ≥ ULN +10 sec). 29.Positive serology for:

1. Hepatitis B: Positive for Hepatitis B surface antigen (HBsAg). Note: Subjects with positive HBsAg but undetectable Hepatitis B virus deoxyribonucleic acid (HBV-DNA) are eligible.
2. Hepatitis C: Positive for Hepatitis C virus (HCV) antibody. Note: Subjects with positive HCV antibody but undetectable HCV ribonucleic acid (HCV-RNA) are eligible.
3. Positive syphilis screening [Treponema pallidum antibody (Tp-Ab)].
4. Known positive history or positive screening for Human Immunodeficiency Virus (HIV).

30.Pregnancy, lactation, or unwillingness to use highly effective contraception from screening until 180 days after last dose.

31.Participation in another investigational drug/device trial within 90 days before screening (excluding vitamin/mineral studies).

32.Uncontrolled major systemic illness at screening; history of stroke, myocardial infarction, or cerebral infarction within 180 days.

33.Major surgery within 1 month before first dose, or presence of unhealed wounds/ulcers/fractures.

34.Any other condition that, in the investigator's opinion, renders the subject unsuitable for trial participation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) Change From Baseline (No. of Letters) to Week 12 | Baseline (Day 0), Week 12

SECONDARY OUTCOMES:
Proportion of subjects who gained at least 5,10 and 15 letters and lose 15 letters baseline to week 12,week 24 and week 52 | Baseline (Day 0), Week 12, Week 24, Week 52
Change From Baseline in CRT(central retina thickness) by visit | Baseline (Day 0), Week 12, Week 24, Week 52
Change from baseline in CNV area from baseline to week 12 and week 52 | Baseline (Day 0), Week 12, Week 52
BCVA Change From Baseline by visit | Baseline (Day 0), Week 24, Week 52
Incidence of drug-related ocular and systemic adverse reactions at Week 12, Week 24, and Week 52. | Baseline (Day 0), Week 12, Week 24, Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No